CLINICAL TRIAL: NCT02078778
Title: Central and Peripheral 24-h Blood Pressure Monitoring in Patients With Hypertension and Obstructive Sleep Apnea Before and After Treatment With Continuous Positive Airway Pressure.
Brief Title: Central and Peripheral Blood Pressure in Treatment of Obstructive Sleep Apnea.
Acronym: HOSI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erling Bjerregaard Pedersen (Other)
Responsible Party: Sponsor-Investigator, Erling Bjerregaard Pedersen, professor, Regional Hospital Holstebro
Organization: Regional Hospital Holstebro (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGH-4-2013; M-2013-304-13 (Other: The Regional Committee of Health Research Ethics)
Record Dates: First submitted 2014-03-01; First posted 2014-03-05 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Hypertension; Obstructive Sleep Apnea
Keywords: Continuous airway pressure; Hypertension; Obstructive sleep apnea
MeSH Terms: conditions — Hypertension; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Patients with hypertension and moderate to severe OSA is treated with CPAP for 3 months.
  Interventions: Device: CPAP

INTERVENTIONS:
Device: CPAP — 3 months of CPAP treatment
  Other Names: S9 AutoSet frem ResMed/MAribo Medico; or; REMstar Auto A-Flex frem Phillips/Respirsonics

SUMMARY:
The purpose of this study is to examine the effect on blood pressure of 3 months of treatment with continuous positive airway pressure (CPAP) in patients with obstructive sleep apnea (OSA).

Hypothesis:

1. Central 24-h blood pressure (BP) monitoring hedges day fluctuations in blood pressure more accurately than peripheral 24-h BP monitoring, because the measurement is painless and does not interfere with the patient / subject's activities during the daytime or nighttime sleep.
2. Blood pressure is elevated in patients with OSA and falls during treatment with CPAP.

3. The renal treatment of salt and water is abnormal in OSA, improved during treatment with CPAP.

4. Quality of life improves during treatment with CPAP

DETAILED DESCRIPTION:
Approximately 20 patients with hypertension and moderate to severe OSA are treated with CPAP 3 months to examine the treatment effect on blood pressure throughout the day, but especially nocturnal, renal treatment of salt and water, and quality of life.

Before and after 3 months of CPAP treatment is made central and peripheral 24-h ambulatory blood pressure monitoring, 24-h urine collection and blood samples.

ELIGIBILITY:
Inclusion Criteria:

* chronic kidney disease (CKD stage I and II), eGFR 60-90 ml/min/1.73 m2 or eGFR> 90 ml/min/1.73 m2 and proteinuria or other signs of kidney damage.
* Obstructive sleep apnea, apnea hypopnea index (AHI) > 15 (moderate to severe)
* Both men and women
* 55-70 years
* Signed consent form

Exclusion Criteria:

* Lack of desire to participate
* Malignant disease
* Abuse of drugs or alcohol
* Pregnant and breastfeeding
* Incompensated heart failure
* Atrial fibrillation
* Liver disease (Alanine aminotransferase (ALT) > 200)
* Severe chronic obstructive pulmonary disease (Forced expiratory volume in 1 second <50% predicted)
* Blood pressure difference between the right and left arm> 10/10 mmHg

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
difference in systolic peripheral BP at night | 3 months
  The difference in systolic BP at night by peripheral BP days before and after 3 months of treatment of OSA with CPAP in patients with hypertension.

SECONDARY OUTCOMES:
Difference i central systolic BP | 3 months
  The difference in systolic BP at night in central BP days before and after 3 months of treatment of OSA with CPAP in patients with hypertension.
Difference i BP throughout the day | 3 months
  The difference in systolic BP and diastolic BP throughout the day, in the daytime and in nighttime between measurements with peripheral and central 24-h blood pressure monitoring before and after 3 months of treatment with CPAP.
Correlation between degree of OSA and kidney function on effect of treatment | 3 months
  The correlation between the treatment effect on blood pressure levels on the one hand and the severity of OSA prior to initiation of treatment and renal function as measured by estimated glomerular filtration rate (eGFR) on the other.
urine auquaporine2 (u-AQP2) and urine epithelial Natrium channel (u-ENaC) | 3 months
  Changes in U-AQP2 and u-ENaC in 24-h urine samples before and after 3 month of treatment.
Plasma renin concentration (PRC), plasma angiotensin II (p-AngII), plasma aldosterone (p-Aldo), plasma vasopressin (P-AVP) and plasma endothelin (p-endothelin). | 3 months
  Changes in PRC, p-AngII, p-Aldo. P-AVP and p-endothelin in blood samples before and after 3 month of treatment.
Quality of life | 3 months
  Changes in the quality of life before and after treatment of OSA with CPAP.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medical Research and Medicine, Holstebro Regional Hospital, Holstebro, Holstebro, Denmark